#### Title of research study: Male Couples Research Study (MCAP)

Investigator: Jason W. Mitchell, PhD, MPH

#### Why am I being invited to take part in a research study?

We invite you to take part in a research study because you are currently in an adult same-sex male relationship who lives in the United States. This form is designed to tell you everything you need to think about before you decide to consent (agree) to be in the study or not to be in the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. You can skip any questions that you do not wish to answer. You can print a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. By accepting the content of this form you will not give up any legal rights.

#### What should I know about a research study?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- Participation is voluntary.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

#### Who can I talk to?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team at 305-243-8813 or send us an email at mcapstudy@gmail.com

This research has been reviewed and approved by an Institutional Review Board ("IRB"). You may talk to them at (305) 243-3195 if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

# Why is this research being done?

Our research study, MCAP, aims to determine whether a prevention "toolkit" can help improve male couples improve their relationships while reducing their risk for HIV and other STIs. The data collected from this research study will be used to help further refine the prevention "toolkit" for other male couples.

# Permission to Take Part in a Human Research Study

#### How long will the research last?

We expect that you will be in this research study for approximately 6 months. Specifically, your time involved in the study will be approximately 1-2 hours at the very beginning of the study, 1 hour at the 3-month mark, and another 1 hour at the end of the study at 6 months. Over the course of the 6 months, you may also be asked to complete a few exercises on the study's website, which may take about 1 hour of your time. You will be notified if you were randomly selected to complete these exercises. Finally, you will be compensated for your time.

#### How many people will be studied?

We expect about 200 male couples will be in this research study nationally.

#### What happens if I say yes, I want to be in this research?

If you agree to participate in this study, you will be asked to do the following:

- 1) Register to gain access to the study website and surveys (2 minutes). You will be asked to provide your contact information so we may contact you to send reminders about completing the study's surveys.
- 2) Complete 3 surveys about your relationship: 1 at the beginning of the study, another in 3 months time, and the 3<sup>rd</sup>/ last survey in 6 months from now. Each survey should take about 30 minutes to complete. If you take part in this study, you will receive a \$25 electronic Amazon gift card via email after each survey is completed. This is to compensate you for your time.
- 3) Explore the various sections of the study website, which will include topics related to sexual health.

# What happens if I do not want to be in this research? What happens if I say yes, but I change my mind later?

You can leave the research at any time and it will not be held against you. The data you provided up to this point may be used for research purposes, but your personal information will not be stored nor used.

## Is there any way being in this study could be bad for me?

All study activities are private. We encourage you to complete the surveys and view the study website in an environment where you feel comfortable and have privacy. You can be certain that what you share will be kept strictly confidential. Your name and contact information will be collected for recruitment purposes, and to send you reminders to complete the surveys.

After completion of each survey, you will be given websites to different resources. These websites may be used to learn more about the health of gay and bisexual men as well as same-sex male couples, and how to access related resources. We will give you this to help address any distress you may feel from the surveys, and topics asked. In addition to these risks, this research may hurt you in ways that are unknown. These may be a minor inconvenience to you.

#### Will being in this study help me any way?

We cannot promise any benefits to you or others from your taking part in this research. However, possible benefits include you gaining a better understanding about your relationship and learning about newer methods of HIV prevention.

### Permission to Take Part in a Human Research Study

Page 3 of 3

#### What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study, to people who have a need to review this information. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB and other representatives of this organization.

All research data will be kept in a secure location. Data will not contain any identifying information, including names.

Certain offices and people may look at study records. University of Miami employees overseeing proper study conduct may look at your study records. These offices include the Office for Human Research Protections, the funder, the University of Miami Miller School of Medicine Institutional Review Board, and the University of Miami Office of Research Compliance. We will keep all records private to the extent we are required to do so by law, even if you admit to illegal activity, with the exception of any reported child and elderly abuse (these instances must be reported). We will not collect any information that will identify you personally for the study. We will not highlight other facts that might point to you when we present this study or publish its results.

#### Can I be removed from the research without my OK?

The person in charge of the research study or the sponsor can remove you from the research study without your approval.

#### What else do I need to know?

This research is being funded by the National Institute of Mental Health.

Do you agree to these terms and wish to participate in this research study? .

"Yes – I agree and wish to participate. You may contact me." X

"No – I do not agree and do not wish to participate." X

Document Revision Date: June 23, 2015